CLINICAL TRIAL: NCT01345240
Title: Immunogenicity of the Hepatitis B Antigen of the GSK Biologicals' Candidate Malaria Vaccine (257049)
Brief Title: Study to Evaluate Immunogenicity of the Hepatitis B Antigen of the GSK Biologicals' Candidate Malaria Vaccine (257049)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113681; 2011-001508-37 (EudraCT Number)
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Malaria; Malaria Vaccines
Keywords: Africa; Plasmodium falciparum; Malaria vaccine; hepatitis B; EPI
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Hepatitis B | interventions — halofantrine; Measles Vaccine; Yellow Fever Vaccine

ARMS (11):
- RTS,S Regimen A Lot 1 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen A, with the RTS,S vaccine administered in its Lot 1 formulation. This RTS,S Vaccination Regimen A included 3 doses of RTS,S vaccine, Lot 1, co-administered with Infanrix™-Hib, Polio Sabin™ and Synflorix™, at Weeks 0, 4 and 8, and 2 doses of Rotarix™ vaccine, at Weeks 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- RTS,S Regimen A Lot 2 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen A, with the RTS,S vaccine administered in its Lot 2 formulation. This RTS,S Vaccination Regimen A included 3 doses of RTS,S vaccine, Lot 2, co-administered with Infanrix™-Hib, Polio Sabin™ and Synflorix™, at Weeks 0, 4 and 8, and 2 doses of Rotarix™ vaccine, at Weeks 6 and 10. In addition, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- RTS,S Regimen A Lot 3 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen A, with the RTS,S vaccine administered in its Lot 3 formulation. This RTS,S Vaccination Regimen A included 3 doses of RTS,S vaccine, Lot 3, co-administered with Infanrix™-Hib, Polio Sabin™ and Synflorix™, at Weeks 0, 4 and 8, and 2 doses of Rotarix™ vaccine, at Weeks 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- RTS,S Regimen B Lot 1 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen B, with the RTS,S vaccine administered in its Lot 1 formulation. This RTS,S Vaccination Regimen B included 3 doses of RTS,S vaccine, Lot 1, co-administered with Infanrix™-Hib and Polio Sabin™, at Weeks 0, 4 and 8, 2 doses of Rotarix™, at Weeks 4 and 8, and 3 doses of Synflorix™ at Weeks 2, 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- RTS,S Regimen B Lot 2 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen B, with the RTS,S vaccine administered in its Lot 2 formulation. This RTS,S Vaccination Regimen B included 3 doses of RTS,S vaccine, Lot 2, co-administered with Infanrix™-Hib and Polio Sabin™, at Weeks 0, 4 and 8, 2 doses of Rotarix™, at Weeks 4 and 8, and 3 doses of Synflorix™ at Weeks 2, 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- RTS,S Regimen B Lot 3 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen B, with the RTS,S vaccine administered in its Lot 3 formulation. This RTS,S Vaccination Regimen B included 3 doses of RTS,S vaccine, Lot 3, co-administered with Infanrix™-Hib and Polio Sabin™, at Weeks 0, 4 and 8, 2 doses of Rotarix™, at Weeks 4 and 8, and 3 doses of Synflorix™ at Weeks 2, 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- RTS,S Regimen C Lot 1 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen C, with the RTS,S vaccine administered in its Lot 1 formulation. This RTS,S Vaccination Regimen C included 3 doses of RTS,S vaccine, Lot 1, co-administered with Infanrix™-Hib and Polio Sabin™, at Weeks 0, 4 and 8, 2 doses of Rotarix™, at Weeks 6 and 10, and 3 doses of Synflorix™ at Weeks 2, 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- RTS,S Regimen C Lot 2 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen C, with the RTS,S vaccine administered in its Lot 2 formulation. This RTS,S Vaccination Regimen C included 3 doses of RTS,S vaccine, Lot 2, co-administered with Infanrix™-Hib and Polio Sabin™, at Weeks 0, 4 and 8, 2 doses of Rotarix™, at Weeks 6 and 10, and 3 doses of Synflorix™ at Weeks 2, 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- RTS,S Regimen C Lot 3 Group (Experimental): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the RTS,S Vaccination Regimen C, with the RTS,S vaccine administered in its Lot 3 formulation. This RTS,S Vaccination Regimen C included 3 doses of RTS,S vaccine, Lot 3, co-administered with Infanrix™-Hib and Polio Sabin™, at Weeks 0, 4 and 8, 2 doses of Rotarix™, at Weeks 6 and 10, and 3 doses of Synflorix™ at Weeks 2, 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. The RTS,S vaccine and Engerix B™ were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049; Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- Engerix B Regimen A Group (Active Comparator): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the Engerix-B Vaccination Regimen A. This regimen included 3 doses of Engerix B™ co-administered with Infanrix™-Hib, Polio Sabin™ and Synflorix™ at Weeks 0, 4 and 8, and 2 doses of Rotarix™, at Weeks 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. Engerix B™ was administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine
- Engerix B Regimen B Group (Active Comparator): Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the Engerix-B Vaccination Regimen B. This regimen included 3 doses of Engerix B™ co-administered with Infanrix™-Hib and Polio Sabin™, at Weeks 0, 4 and 8, 2 doses of Rotarix™ vaccine, at Weeks 4 and 8, and 3 doses of Synflorix™ at Weeks 2, 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix™-Hib and Synflorix™, at Month 16, and one booster dose of Engerix B™ vaccine, at Month 50. Engerix B™ was administered intramuscularly (IM) in the left anterolateral thigh, Infanrix™-Hib IM in the right deltoid, Synflorix™ IM in the right anterolateral thigh, and Rotarix™ and Polio Sabin™ orally. The measles and yellow fever vaccines were administered IM in the deltoid.
  Interventions: Biological: Engerix-B™ vaccine; Biological: Infanrix/Hib™ vaccine; Biological: Polio Sabin™ vaccine; Biological: Rotarix™ vaccine; Biological: Synflorix™ vaccine; Biological: Measles vaccine; Biological: Yellow fever vaccine

INTERVENTIONS:
Biological: GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine 257049 — Children enrolled in 9 groups will receive 3 doses of the candidate malaria vaccine (Lot 1, 2 and 3) by intramuscular injection.
  Arms: RTS,S Regimen A Lot 1 Group; RTS,S Regimen A Lot 2 Group; RTS,S Regimen A Lot 3 Group; RTS,S Regimen B Lot 1 Group; RTS,S Regimen B Lot 2 Group; RTS,S Regimen B Lot 3 Group; RTS,S Regimen C Lot 1 Group; RTS,S Regimen C Lot 2 Group; RTS,S Regimen C Lot 3 Group
Biological: Engerix-B™ vaccine — Children enrolled in 2 groups will receive 4 doses of Engerix-B™ vaccine by intramuscular injection. Children enrolled in all other groups will receive one dose of Engerix-B vaccine by intramuscular injection.
Biological: Infanrix/Hib™ vaccine — Children enrolled in all 11 groups will receive 4 doses of Infanrix/Hib™ vaccine by intramuscular injection
Biological: Polio Sabin™ vaccine — Children enrolled in all 11 groups will receive 3 doses of Polio Sabin™ by intramuscular injection.
Biological: Rotarix™ vaccine — Children enrolled in all 11 groups will receive 2 doses of oral Rotarix™ vaccine.
Biological: Synflorix™ vaccine — Children enrolled in all 11 groups will receive 4 doses of Synflorix™ vaccine by intramuscular injection.
Biological: Measles vaccine — Children enrolled in all 11 groups will receive 1 dose of measles vaccine by intramuscular injection.
Biological: Yellow fever vaccine — Children enrolled in all 11 groups will receive 1 dose of yellow fever vaccine by intramuscular injection.

SUMMARY:
This study has been designed to support the indication of the candidate vaccine (also referred to as GSK 257049 or RTS,S in this record) against hepatitis B virus infection, when administered as a primary vaccination integrated into an Expanded Program on Immunization (EPI) regimen to infants living in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* A male or female infant aged between 8 and 12 weeks inclusive at the time of first vaccination
* Signed or thumb-printed informed consent obtained from the parent(s)/Legally Acceptable Representative [LAR(s)] of the child. Where parent(s)/LAR(s) are illiterate, the consent form will be countersigned by an independent witness
* Subjects who the investigator believes that their parent(s)/LAR(s) can and will comply with the requirements of the protocol
* Healthy subjects as established by medical history and clinical examination before entering into the study
* Born to a mother who is Hepatitis B surface antigen (HBsAg) negative
* Born to a mother who is Human Immunodeficiency Virus (HIV) negative
* Born after a normal gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Child in care
* Acute disease and/or fever at the time of enrolment
* Serious acute or chronic illness determined by clinical or physical examination and laboratory screening tests
* Laboratory screening tests out of range
* Previous vaccination with diphtheria, tetanus, pertussis, Haemophilus influenzae type b, Streptococcus pneumoniae, hepatitis B vaccine or rotavirus vaccines.
* Planned administration/administration of a licensed vaccine not foreseen by the study protocol within 7 days of the first dose of study vaccine.
* Use of a drug or vaccine that is not approved for that indication other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins and/or any blood products in the period between birth and Dose 1 and within the three months preceding planned vaccine administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs in the period between birth and Dose 1.
* Concurrently participating in another clinical study at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Same sex twin
* Maternal death
* History of allergic reactions or anaphylaxis to previous immunizations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.
* Any other findings that the investigator feels would result in data collected being incomplete or of poor quality.
* Previous participation in any other malaria vaccine trial.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 705 (Actual)
Dates: Start 2011-11-17 (Actual); Primary Completion 2013-01-09 (Actual); Study Completion 2017-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Ouagadougou, Burkina Faso
- GSK Investigational Site, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Valea I, Adjei S, Usuf E, Traore O, Ansong D, Tinto H, Owusu Boateng H, Leach A, Mwinessobaonfou Some A, Buabeng P, Vekemans J, Nana LA, Kotey A, Vandoolaeghe P, Ouedraogo F, Sambian D, Lievens M, Tahita MC, Rettig T, Jongert E, Lompo P, Idriss A, Borys D, Ouedraogo S, Prempeh F, Habib MA, Schuerman L, Sorgho H, Agbenyega T. Immune response to the hepatitis B antigen in the RTS,S/AS01 malaria vaccine, and co-administration with pneumococcal conjugate and rotavirus vaccines in African children: A randomized controlled trial. Hum Vaccin Immunother. 2018 Jun 3;14(6):1489-1500. doi: 10.1080/21645515.2018.1442996. Epub 2018 Apr 13. PMID 29630438
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 4 phases, a Primary Vaccination Phase (up to Month (M) 3), a Safety Follow-Up Phase (M3-8), a First Immunogenicity Follow-Up (FU) Phase (M8-26), and a Second Immunogenicity FU Phase (M26 to study end at M51).
Groups:
- RTS,S Regimen A Group: This group results from the pooling of the RTS,S Regimen A Lot 1, RTS,S Regimen A Lot 2 and RTS,S Regimen A Lot 3 groups. Subjects, healthy male and female infants aged between 8 and 12 weeks inclusive at the time of first vaccination, received 3 doses of RTS,S vaccine, Lot 1, 2 or 3, co-administered with Infanrix-Hib, Polio Sabin and Synflorix, at Weeks 0, 4 and 8, and 2 doses of Rotarix vaccine, at Weeks 6 and 10. In addition, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix-Hib and Synflorix, at Month 16, and one booster dose of Engerix B vaccine, at Month 50. The RTS,S vaccine and Engerix B were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
- RTS,S Regimen B Group: This group results from the pooling of the RTS,S Regimen B Lot 1, RTS,S Regimen B Lot 2 and RTS,S Regimen B Lot 3 groups. Subjects, healthy male and female infants aged between 8 and 12 weeks inclusive at the time of first vaccination, received 3 doses of RTS,S vaccine, Lot 1, 2 or 3, co-administered with Infanrix-Hib and Polio Sabin, at Weeks 0, 4 and 8, 2 doses of Rotarix, at Weeks 4 and 8, and 3 doses of Synflorix at Weeks 2, 6 and 10. In addition, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix-Hib and Synflorix, at Month 16, and one booster dose of Engerix B vaccine, at Month 50. The RTS,S vaccine and Engerix B were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
- RTS,S Regimen C Group: This group results from the pooling of the RTS,S Regimen C Lot 1, RTS,S Regimen C Lot 2 and RTS,S Regimen C Lot 3 groups. Subjects, healthy male and female infants aged between 8 and 12 weeks inclusive at the time of first vaccination, received 3 doses of RTS,S vaccine, Lot 1, 2 or 3, co-administered with Infanrix-Hib and Polio Sabin, at Weeks 0, 4 and 8, 2 doses of Rotarix, at Weeks 6 and 10, and 3 doses of Synflorix at Weeks 2, 6 and 10. In addition, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix-Hib and Synflorix, at Month 16, and one booster dose of Engerix B vaccine, at Month 50. The RTS,S vaccine and Engerix B were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
- Engerix B Regimen A Group: Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the Engerix-B Vaccination Regimen A. This regimen included 3 doses of Engerix B co-administered with Infanrix-Hib, Polio Sabin and Synflorix at Weeks 0, 4 and 8, and 2 doses of Rotarix, at Weeks 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix-Hib and Synflorix, at Month 16, and one booster dose of Engerix B vaccine, at Month 50. Engerix B was administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
- Engerix B Regimen B Group: Subjects, healthy male and female infants between 8 and 12 weeks of age inclusive at the time of first vaccination, received the Engerix-B Vaccination Regimen B. This regimen included 3 doses of Engerix B co-administered with Infanrix-Hib and Polio Sabin, at Weeks 0, 4 and 8, 2 doses of Rotarix vaccine, at Weeks 4 and 8, and 3 doses of Synflorix at Weeks 2, 6 and 10. Additionally, subjects also received one dose of vaccine against yellow fever and against measles, at Week 32, and one booster dose of Infanrix-Hib and Synflorix, at Month 16, and one booster dose of Engerix B vaccine, at Month 50. Engerix B was administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
Period: Overall Study
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Started | 142 | 142 | 141 | 141 | 139
Completed | 131 | 128 | 123 | 132 | 129
Not Completed | 11 | 14 | 18 | 9 | 10
Not completed — Adverse Event | 3 | 5 | 4 | 2 | 1
Not completed — Lost to Follow-up | 8 | 9 | 14 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group | Total
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139 | 705
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.4 (0.83) | 8.3 (0.62) | 8.3 (0.69) | 8.3 (0.74) | 8.3 (0.74) | 8.32 (0.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 69 | 67 | 81 | 63 | 339
  Male | 83 | 73 | 74 | 60 | 76 | 366
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage/African American | 142 | 142 | 141 | 141 | 139 | 705

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Seroprotected Subjects Against Anti-Hepatitis B (HBs) Antigen
Description: A seroprotected subject was defined as a subject with anti-HBs antibody titers greater than or equal to (>=) the cut-off of 10 mili-international units per mililiter (mIU/mL). A decrease in the specificity of the anti-HBs ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete retesting/reanalysis, with study groups pooled by primary vaccine administered (RTS,S vs Engerix -B).
Time Frame: At Month 3, aka at one month post Dose 3 of RTS,S vaccine or Engerix-B
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity measures were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- RTS,S Group: Subjects in this group were subjects from the RTS,S Regimen A, RTS,S Regimen B, and RTS,S Regimen C groups who were administered a 3-dose primary vaccination course of the RTS,S vaccine in any of its formulations, Lot 1, 2 or 3, at Weeks 0, 4 and 8. Subjects in this group were also administered, according to varied schedules depending on the RTS,S vaccination regimen received, doses of Infanrix-Hib, Polio Sabin, Rotarix, Synflorix, Rotarix, Engerix B and vaccines against yellow fever and against measles. The RTS,S vaccine and Engerix B were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
- Engerix B Group: Subjects in this group were subjects from the Engerix B Regimen A and Engerix B Regimen B groups who were administered Engerix B as a 3-dose primary vaccination course, at Weeks 0, 4 and 8, followed by a booster dose, at Month 50. Subjects in this group were also administered, according to varied schedules, depending on the vaccination regimen they were allocated too in their respective group, doses Infanrix-Hib, Polio Sabin, Rotarix, Synflorix, Rotarix and of vaccines against yellow fever and against measles. Engerix B was administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
Arm/Group | RTS,S Group | Engerix B Group
Number analyzed (Participants) | 397 | 253
Percentage of subjects | 100 [99.1 to 100] | 96 [92.9 to 98.1]
Statistical Analysis 1: Comparison: RTS,S Group vs Engerix B Group; Non-inferiority of the immune response to the hepatitis B antigen induced by RTS,S/AS01E vaccine versus a licensed hepatitis B vaccine; Test type: Non-Inferiority — Criteria for non-inferiority: one month post Dose 3, upper limit (UL) of the 2-sided 95% confidence interval (CI) on the difference in percent seroprotection below 5% between recipients of licensed hepatitis B vaccine (Engerix-B) and recipients of RTS,S/AS01E vaccine; Difference in percent seroprotection = -3.95, 95% CI 2-sided [-7.12 to -2.16]

2. Primary Outcome: Anti-Hepatitis B (HBs) Antibody Concentrations for RTS,S Group and Engerix B Group
Description: Concentrations, by enzyme-linked immunosorbent assay (ELISA), were presented as geometric mean concentrations (GMCs), and expressed in milli-international units per milliliter (mIU/mL). The assay cut-off was the seropositivity cut-off value of greater than or equal to (>=) 10 mIU/mL. A decrease in the specificity of the anti-HBs ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete retesting/reanalysis, with study groups pooled by primary vaccine administered (RTS,S vs Engerix-B).
Time Frame: At Month 3, aka at one month post Dose 3 of RTS,S vaccine or Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RTS,S Group | Engerix B Group
Number analyzed (Participants) | 397 | 253
mIU/mL | 6412.7 [5732.9 to 7173.0] | 377.4 [310.6 to 458.7]

3. Primary Outcome: Anti-Hepatitis B (HBs) Antibody Concentrations for All Study Groups
Description: Concentrations, by enzyme-linked immunosorbent assay (ELISA), were presented as geometric mean concentrations (GMCs), and expressed in milli-international units per milliliter (mIU/mL). The assay cut-off was the seropositivity cut-off value of greater than or equal to (>=) 10 mIU/mL. A decrease in the specificity of the anti-HBs ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete retesting/reanalysis, for each RTS,S Regimen A, B, C and each Engerix B Regimen A and B study groups.
Time Frame: At Month 3, aka at one month post Dose 3 of RTS,S vaccine or Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 140 | 123 | 134 | 135 | 118
mIU/mL | 5467.6 [4493.8 to 6652.5] | 6989.9 [5747.5 to 8501.0] | 6998.7 [5779.1 to 8475.7] | 334.4 [253.4 to 441.4] | 433.4 [329.5 to 570.1]

4. Secondary Outcome: Anti-Hepatitis B (HBs) Antibody Concentrations at Month 3
Description: Concentrations, by enzyme-linked immunosorbent assay (ELISA), were presented as geometric mean concentrations (GMCs), and expressed in milli-international units per milliliter (mIU/mL). The assay cut-off was the seropositivity cut-off value of greater than or equal to (>=) 10 mIU/mL. A decrease in the specificity of the anti-HBs ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete retesting/reanalysis. Results presented are for the study groups receiving the RTS,S vaccine, pooled by vaccine lot, that is, for the RTS,S Lot 1, RTS,S Lot 2, and RTS,S Lot 3 groups, as defined below.
Time Frame: At Month 3, aka at one month post Dose 3 of RTS,S vaccine or Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- RTS,S Lot 1 Group: Subjects in this group were subjects from the RTS,S Regimen A, RTS,S Regimen B, and RTS,S Regimen C groups who were administered a 3-dose primary vaccination course of the RTS,S vaccine in its Lot 1 formulation only, at Weeks 0, 4 and 8. Subjects in this group were also administered, according to varied schedules depending on the RTS,S vaccination regiment received, doses of Infanrix-Hib, Polio Sabin, Rotarix, Synflorix, Rotarix, Engerix B and vaccines against yellow fever and against measles. The RTS,S vaccine and Engerix B were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
- RTS,S Lot 2 Group: Subjects in this group were subjects from the RTS,S Regimen A, RTS,S Regimen B, and RTS,S Regimen C groups who were administered a 3-dose primary vaccination course of the RTS,S vaccine in its Lot 2 formulation only, at Weeks 0, 4 and 8. Subjects in this group were also administered, according to varied schedules depending on the RTS,S vaccination regiment received, doses of Infanrix-Hib, Polio Sabin, Rotarix, Synflorix, Rotarix, Engerix B and vaccines against yellow fever and against measles. The RTS,S vaccine and Engerix B were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
- RTS,S Lot 3 Group: Subjects in this group were subjects from the RTS,S Regimen A, RTS,S Regimen B, and RTS,S Regimen C groups who were administered a 3-dose primary vaccination course of the RTS,S vaccine in its Lot 3 formulation only, at Weeks 0, 4 and 8. Subjects in this group were also administered, according to varied schedules depending on the RTS,S vaccination regimen received, doses of Infanrix-Hib, Polio Sabin, Rotarix, Synflorix, Rotarix, Engerix B and vaccines against yellow fever and against measles. The RTS,S vaccine and Engerix B were administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
Arm/Group | RTS,S Lot 1 Group | RTS,S Lot 2 Group | RTS,S Lot 3 Group
Number analyzed (Participants) | 132 | 134 | 131
mIU/mL | 6214.3 [5115.6 to 7548.9] | 6826.1 [5569.4 to 8366.3] | 6209.2 [5144.2 to 7494.8]
Statistical Analysis 1: Comparison: RTS,S Lot 1 Group vs RTS,S Lot 2 Group; To demonstrate the lot-to-lot consistency in terms of anti-HBs immunogenicity between three commercial lots of the RTS,S/AS01E candidate malaria vaccine; Test type: Equivalence — Criteria for consistency: one month post Dose 3 of RTS,S/AS01E, the two-sided 95% confidence interval (CI) of the geometric mean concentration (GMC) ratio between all pairs of lots are within [0.5, 2]; ANOVA; GMC ratio = 0.91, 95% CI 2-sided [0.69 to 1.20]
Statistical Analysis 2: Comparison: RTS,S Lot 1 Group vs RTS,S Lot 3 Group; [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; ANOVA; GMC ratio = 1.00, 95% CI 2-sided [0.76 to 1.32]
Statistical Analysis 3: Comparison: RTS,S Lot 2 Group vs RTS,S Lot 3 Group; [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; ANOVA; GMC ratio = 1.10, 95% CI 2-sided [0.84 to 1.45]

5. Secondary Outcome: Anti-Hepatitis B (HBs) Antibody Concentrations at Month 14 and 26
Description: Concentrations, by enzyme-linked immunosorbent assay (ELISA), were presented as geometric mean concentrations (GMCs), and expressed in milli-international units per milliliter (mIU/mL). The assay cut-off was the seropositivity cut-off value of greater than or equal to (>=) 10 mIU/mL. A decrease in the specificity of the anti-HBs ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete retesting/reanalysis. Results presented are for each RTS,S Regimen A, B & C, and for each Engerix B Regimen A & B study groups.
Time Frame: At Months 14 and 26, aka at 12 and 24 months post Dose 3 of RTS,S vaccine or Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 133 | 118 | 129 | 127 | 114
mIU/mL
  Anti-HBs - At Month 14 | 1530.1 [1259.4 to 1859.1] | 2430.9 [1975.7 to 2991.0] | 2189.1 [1840.3 to 2603.9] | 119.5 [91.0 to 157.0] | 137.5 [103.3 to 183.2]
  Anti-HBs - At Month 26: number analyzed (Participants) | 132 | 109 | 124 | 125 | 110
  Anti-HBs - At Month 26 | 1092.6 [867.4 to 1376.3] | 1896.0 [1487.2 to 2417.3] | 1849.8 [1478.9 to 2313.6] | 68.8 [50.7 to 93.3] | 71.0 [51.6 to 97.8]

6. Secondary Outcome: Anti-Hepatitis B (HBs) Antibody Concentrations at Month 38, 50 and 51
Description: as for outcome 5
Time Frame: At Months 38, 50 and 51, aka 36 and 48 months post Dose 3 of RTS,S vaccine or Engerix-B and one month post the Month 50 booster dose of Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 131 | 111 | 122 | 127 | 106
mIU/mL
  Month 38: number analyzed (Participants) | 128 | 107 | 120 | 125 | 105
  Month 38 | 706.8 [548.0 to 911.6] | 1081.7 [845.3 to 1384.2] | 977.4 [786.7 to 1214.3] | 39.0 [29.0 to 52.4] | 41.2 [29.8 to 57.0]
  Month 50: number analyzed (Participants) | 128 | 111 | 122 | 127 | 106
  Month 50 | 499.4 [382.2 to 652.6] | 765.3 [590.5 to 992.0] | 807.3 [649.6 to 1003.4] | 29.2 [22.0 to 38.7] | 32.9 [23.9 to 45.4]
  Month 51: number analyzed (Participants) | 131 | 109 | 122 | 124 | 105
  Month 51 | 32345.9 [24758.5 to 42258.4] | 54977.1 [43579.1 to 69356.4] | 59630.0 [48606.1 to 73154.0] | 8995.0 [5935.8 to 13631.0] | 9578.9 [6374.2 to 14395.0]

7. Secondary Outcome: Concentrations of Antibodies to the Hepatitis B RF1 Surface Antigen (Anti-HBs RF1) at Month 3
Description: Anti-HBs RF1 antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and presented as geometric mean concentrations (GMCs) expressed in ELISA units per milliliter (EL.U/mL). The assay cut-off was the seropositivity cut-off value of greater than or equal to (>=) 33 EL.U/mL. The table shows results for each RTS,S Regimen A, B & C, and for each Engerix B Regimen A & B study groups.
Time Frame: At Month 3, aka at one month post Dose 3 of RTS,S vaccine or Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 141 | 123 | 135 | 135 | 117
EL.U/mL | 268.7 [226.8 to 318.3] | 327.1 [272.2 to 393.1] | 335.5 [283.2 to 397.5] | 25.5 [22.8 to 28.7] | 28.7 [24.6 to 33.4]

8. Secondary Outcome: Concentrations of Antibodies to the Hepatitis B RF1 Surface Antigen (Anti-HBs RF1) at Month 51
Description: as for outcome 7
Time Frame: At Month 51, aka one month post the Month 50 booster dose of Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 124 | 104 | 113 | 107 | 95
EL.U/mL | 307.8 [239.0 to 396.4] | 471.6 [372.5 to 597.1] | 514.5 [415.3 to 637.5] | 120.5 [86.6 to 167.6] | 127.9 [94.5 to 173.1]

9. Secondary Outcome: Anti-circumsporozoite Protein (Anti-CS) Antibody Concentrations at Month 3
Description: Anti-CS antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and presented as geometric mean concentrations (GMCs) expressed in ELISA units per milliliter (EL.U/mL). The assay cut-off was the seropositivity cut-off value of greater than or equal to (>=) 0.5 EL.U/mL. The table shows results for each RTS,S Regimen A, B & C, and for each Engerix B Regimen A & B study groups.
Time Frame: At Month 3, aka at one month post Dose 3 of RTS,S vaccine or Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 141 | 123 | 136 | 135 | 118
EL.U/mL | 142.2 [116.4 to 173.7] | 188.5 [156.5 to 227.0] | 205.5 [167.3 to 252.5] | 0.3 [0.3 to 0.3] | 0.3 [0.3 to 0.4]

10. Secondary Outcome: Anti-circumsporozoite Protein (Anti-CS) Antibody Concentrations at Month 14
Description: Anti-CS antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and presented as geometric mean concentrations (GMCs) expressed in ELISA units per milliliter (EL.U/mL). The assay cut-off was the seropositivity cut-off value of greater than or equal to (>=) 0.5 EL.U/mL. The table shows results for each RTS,S Regimen A, B & C, and for each Engerix B Regimen A & B study groups. No anti-CS results are available for the time point 24 months post Dose 3 (Month 26) because the quantity of serum available for the anti-CS assay was insufficient for many samples.
Time Frame: At Month 14, aka at 12 months post Dose 3 of RTS,S vaccine or Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 91 | 82 | 96 | 85 | 76
EL.U/mL | 5.7 [4.2 to 7.7] | 6.8 [5.0 to 9.4] | 7.5 [5.3 to 10.6] | 0.3 [0.3 to 0.3] | 0.3 [0.3 to 0.4]

11. Secondary Outcome: Anti-circumsporozoite Protein (Anti-CS) Antibody Concentrations at Month 38 and 50
Description: Anti-CS antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and presented as geometric mean concentrations (GMCs) expressed in ELISA units per milliliter (EL.U/mL). The assay cut-off was the seropositivity cut-off value of greater than or equal to (>=) 1.9 EL.U/mL. The table shows results for each RTS,S Regimen A, B & C, and for each Engerix B Regimen A & B study groups.
Time Frame: At Months 38 and 50, aka 36 and 48 months post Dose 3 of RTS,S vaccine or Engerix-B
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 131 | 111 | 122 | 127 | 107
EL.U/mL
  Month 38: number analyzed (Participants) | 131 | 107 | 121 | 126 | 106
  Month 38 | 2.6 [2.2 to 3.1] | 2.8 [2.3 to 3.4] | 3.5 [2.9 to 4.2] | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  Month 50: number analyzed (Participants) | 128 | 111 | 122 | 127 | 107
  Month 50 | 2.3 [2.0 to 2.7] | 2.4 [2.0 to 2.8] | 2.7 [2.3 to 3.2] | 1.1 [1.0 to 1.1] | 1.1 [1.0 to 1.3]

12. Secondary Outcome: Pneumococcal Antibody Concentrations Against Synflorix Pneumococcal Vaccine Serotypes at Month 3
Description: Antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), and expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The pneumococcal vaccine serotypes assessed were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The cut-off of the assay, by GSK assay, was greater than or equal to (>=) 0.2 µg/mL. This corresponds to the standard ELISA value of 0.35 μg/mL. This outcome concerns the subjects who received the RTS,S or Engerix-B vaccine co-administered with Synflorix. Results presented are for the study groups pooled by co-administration, that is, for the RTS,S Regimen A and Engerix-B Regimen A groups.
Time Frame: At Month 3, aka at one month post Dose 3 of Synflorix
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | RTS,S Regimen A Group | Engerix B Regimen A Group
Number analyzed (Participants) | 141 | 135
µg/mL
  ANTI-1 | 3.1 [2.8 to 3.6] | 3.6 [3.1 to 4.2]
  ANTI-4: number analyzed (Participants) | 141 | 134
  ANTI-4 | 3.5 [3.0 to 4.0] | 4.2 [3.5 to 4.9]
  ANTI-5 | 5.1 [4.5 to 5.8] | 6.5 [5.6 to 7.4]
  ANTI-6B | 1.1 [0.8 to 1.3] | 1.2 [1.0 to 1.6]
  ANTI-7F | 4.4 [3.9 to 4.9] | 4.9 [4.3 to 5.7]
  ANTI-9V | 2.8 [2.4 to 3.3] | 3.7 [3.3 to 4.2]
  ANTI-14: number analyzed (Participants) | 141 | 134
  ANTI-14 | 5.8 [5.0 to 6.7] | 5.7 [4.7 to 7.0]
  ANTI-18C: number analyzed (Participants) | 141 | 134
  ANTI-18C | 3.4 [2.8 to 4.1] | 6.2 [5.1 to 7.5]
  ANTI-19F: number analyzed (Participants) | 141 | 134
  ANTI-19F | 4.2 [3.4 to 5.2] | 5.1 [4.1 to 6.4]
  ANTI-23F: number analyzed (Participants) | 140 | 134
  ANTI-23F | 1.3 [1.1 to 1.6] | 1.5 [1.1 to 1.9]
Statistical Analysis 1: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against serotype 1 responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — Criteria for non-inferiority: one month post Dose 3, upper limit (UL) of the 2-sided 95% confidence interval (CI) on the GMC ratios of 10 pneumococcal serotypes titers (measured with an ELISA test), is below a limit of 2 for the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E; ANOVA; GMC ratio = 1.15, 95% CI 2-sided [0.95 to 1.39]
Statistical Analysis 2: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against serotype 4 responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 1.20, 95% CI 2-sided [0.97 to 1.48]
Statistical Analysis 3: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against serotype 5 responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 1.27, 95% CI 2-sided [1.06 to 1.52]
Statistical Analysis 4: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against serotype 6B responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 1.17, 95% CI 2-sided [0.83 to 1.65]
Statistical Analysis 5: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against serotype 7F responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 1.12, 95% CI 2-sided [0.94 to 1.33]
Statistical Analysis 6: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against serotype 9V responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 1.32, 95% CI 2-sided [1.08 to 1.63]
Statistical Analysis 7: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against serotype 14 responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 0.99, 95% CI 2-sided [0.77 to 1.27]
Statistical Analysis 8: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against 18C responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 1.81, 95% CI 2-sided [1.38 to 2.38]
Statistical Analysis 9: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against serotype 19F responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 1.21, 95% CI 2-sided [0.89 to 1.65]
Statistical Analysis 10: Comparison: RTS,S Regimen A Group vs Engerix B Regimen A Group; To demonstrate the non-inferiority of antibody against 23F responses to the pneumococcal conjugate vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; ANOVA; GMC ratio = 1.12, 95% CI 2-sided [0.81 to 1.55]

13. Secondary Outcome: Pneumococcal Antibody Concentrations Against Synflorix Pneumococcal Vaccine Serotypes at Month 17
Description: Antibody concentrations were measured by GSK assay, and expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The pneumococcal vaccine serotypes assessed were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. The cut-off of the assay, by GSK assay, was greater than or equal to (>=) 0.2 μg/mL. This corresponds to the standard ELISA value of 0.35 μg/mL. This outcome concerns the subjects who received the RTS,S or Engerix -B vaccine co-administered with Synflorix. Results presented are for the study groups pooled by co-administration, that is, for the RTS,S Regimen A and Engerix -B Regimen A groups.
Time Frame: At Month 17, aka one month post the Month 16 booster dose of Synflorix
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | RTS,S Regimen A Group | Engerix B Regimen A Group
Number analyzed (Participants) | 133 | 126
μg/mL
  ANTI-1 | 4.5 [3.8 to 5.4] | 5.4 [4.5 to 6.4]
  ANTI-4: number analyzed (Participants) | 132 | 125
  ANTI-4 | 6.1 [5.1 to 7.2] | 6.8 [5.7 to 8.0]
  ANTI-5 | 6.5 [5.5 to 7.8] | 7.6 [6.4 to 9.1]
  ANTI-6B | 4.7 [4.0 to 5.5] | 4.1 [3.5 to 4.9]
  ANTI-7F | 7.1 [6.2 to 8.2] | 7.2 [6.3 to 8.2]
  ANTI-9V | 6.0 [5.1 to 7.1] | 5.7 [4.9 to 6.6]
  ANTI-14 | 9.0 [7.6 to 10.7] | 9.0 [7.4 to 10.8]
  ANTI-18C | 13.7 [11.5 to 16.3] | 14.5 [12.3 to 17.2]
  ANTI-19F | 6.0 [4.9 to 7.4] | 7.2 [5.8 to 8.8]
  ANTI-23F | 4.1 [3.4 to 5.1] | 3.9 [3.2 to 4.8]

14. Secondary Outcome: Titers for Opsonophagocytic Activity Against Synflorix Pneumococcal Vaccine Serotypes at Month 3
Description: The pneumococcal vaccine serotypes assessed were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Streptococcus pneumoniae opsonophagocytic activity was presented as the dilution of serum (opsonic titer) able to sustain 50 % killing of live pneumococci under the assay conditions, expressed as geometric mean titers (GMTs). The cut-off of the assay was an opsonic dilution >= 8. This outcome concerns the subjects who received the RTS,S or Engerix-B vaccine co-administered with Synflorix. Results presented are for the study groups pooled by co-administration, that is, for the RTS,S Regimen A and Engerix-B Regimen A groups.
Time Frame: At Month 3, aka at one month (1M) post Dose 3 of Synflorix
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RTS,S Regimen A Group | Engerix B Regimen A Group
Number analyzed (Participants) | 133 | 124
Titer
  OPSONO-1: number analyzed (Participants) | 132 | 124
  OPSONO-1 | 48.9 [34.6 to 68.9] | 65.0 [45.0 to 93.7]
  OPSONO-4: number analyzed (Participants) | 130 | 123
  OPSONO-4 | 768.3 [617.6 to 955.8] | 810.9 [676.5 to 972.0]
  OPSONO-5 | 77.6 [61.9 to 97.3] | 93.8 [73.6 to 119.6]
  OPSONO-6B: number analyzed (Participants) | 128 | 121
  OPSONO-6B | 444.4 [295.0 to 669.5] | 389.3 [250.1 to 606.1]
  OPSONO-7F: number analyzed (Participants) | 132 | 124
  OPSONO-7F | 3774.0 [3232.7 to 4405.8] | 3947.4 [3338.3 to 4667.7]
  OPSONO-9V: number analyzed (Participants) | 132 | 122
  OPSONO-9V | 1257.7 [977.3 to 1618.7] | 1469.3 [1180.4 to 1828.8]
  OPSONO-14: number analyzed (Participants) | 132 | 123
  OPSONO-14 | 1426.3 [1136.0 to 1790.9] | 1269.0 [965.1 to 1668.6]
  OPSONO-18C: number analyzed (Participants) | 124 | 118
  OPSONO-18C | 192.6 [139.2 to 266.4] | 249.7 [185.0 to 337.0]
  OPSONO-19F: number analyzed (Participants) | 129 | 123
  OPSONO-19F | 159.3 [109.9 to 231.0] | 228.8 [160.4 to 326.3]
  OPSONO-23F: number analyzed (Participants) | 132 | 121
  OPSONO-23F | 760.9 [476.3 to 1215.5] | 735.6 [456.3 to 1185.9]

15. Secondary Outcome: Titers for Opsonophagocytic Activity Against Synflorix Pneumococcal Vaccine Serotypes at Month 17
Description: The pneumococcal vaccine serotypes assessed were the serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Streptococcus pneumoniae opsonophagocytic activity was presented as the dilution of serum (opsonic titer) able to sustain 50 % killing of live pneumococci under the assay conditions, expressed as geometric mean titers (GMTs). The cut-off of the assay was an opsonic dilution >= 8. This outcome concerns the subjects who received the RTS,S or Engerix -B vaccine co-administered with Synflorix . Results presented are for the study groups pooled by co-administration, that is, for the RTS,S Regimen A and Engerix -B Regimen A groups.
Time Frame: At Month 17, aka one month post the Month 16 booster dose of Synflorix
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RTS,S Regimen A Group | Engerix B Regimen A Group
Number analyzed (Participants) | 130 | 121
Titer
  OPSONO-1 | 649.9 [464.7 to 908.9] | 840.1 [603.4 to 1169.7]
  OPSONO-4: number analyzed (Participants) | 126 | 116
  OPSONO-4 | 2347.1 [1847.4 to 2982.0] | 2527.8 [2064.1 to 3095.7]
  OPSONO-5: number analyzed (Participants) | 129 | 121
  OPSONO-5 | 324.2 [244.1 to 430.5] | 392.8 [291.3 to 529.6]
  OPSONO-6B: number analyzed (Participants) | 130 | 116
  OPSONO-6B | 955.3 [761.4 to 1198.6] | 828.2 [652.7 to 1050.9]
  OPSONO-7F: number analyzed (Participants) | 130 | 118
  OPSONO-7F | 9167.3 [7979.2 to 10532.3] | 7794.6 [6577.6 to 9236.8]
  OPSONO-9V: number analyzed (Participants) | 130 | 118
  OPSONO-9V | 3035.3 [2523.3 to 3651.3] | 3164.6 [2669.8 to 3751.1]
  OPSONO-14: number analyzed (Participants) | 127 | 119
  OPSONO-14 | 1975.7 [1565.8 to 2493.0] | 1865.0 [1463.9 to 2375.9]
  OPSONO-18C: number analyzed (Participants) | 127 | 115
  OPSONO-18C | 1694.1 [1188.6 to 2414.7] | 1548.7 [1096.3 to 2188.0]
  OPSONO-19F | 344.5 [223.0 to 532.3] | 469.7 [320.0 to 689.4]
  OPSONO-23F: number analyzed (Participants) | 127 | 118
  OPSONO-23F | 3199.8 [2543.7 to 4025.1] | 3198.1 [2526.5 to 4048.4]

16. Secondary Outcome: Anti-protein D (PD) Antibody Concentrations at Month 3
Description: Anti-PD antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs), in ELISA units per milliliter (EL.U/mL). The cut-off of the assay was the seropositivity cut-off value of greater than or equal to 100 EL.U/mL. This outcome concerns the subjects who received the RTS,S or Engerix-B vaccine co-administered with Synflorix. Results presented are for the study groups pooled by co-administration, that is, for the RTS,S Regimen A and Engerix-B Regimen A groups.
Time Frame: At Month 3, aka at one month post Dose 3 of Synflorix
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Regimen A Group | Engerix B Regimen A Group
Number analyzed (Participants) | 141 | 134
EL.U/mL | 2435.3 [2204.3 to 2690.6] | 2956.7 [2647.5 to 3302.1]

17. Secondary Outcome: Anti-protein D (PD) Antibody Concentrations at Month 17
Description: Anti-PD antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs), in ELISA units per milliliter (EL.U/mL). The cut-off of the assay was the seropositivity cut-off value of greater than or equal to 100 EL.U/mL. This outcome concerns the subjects who received the RTS,S or Engerix -B vaccine co-administered with Synflorix. Results presented are for the study groups pooled by co-administration, that is, for the RTS,S Regimen A and Engerix -B Regimen A groups.
Time Frame: At Month 17, aka one month post the Month 16 booster dose of Synflorix
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Regimen A Group | Engerix B Regimen A Group
Number analyzed (Participants) | 133 | 126
EL.U/mL | 2648.3 [2194.2 to 3196.4] | 2819.1 [2391.1 to 3323.7]

18. Secondary Outcome: Concentrations of Antibodies Against Acellular B-pertussis (BPT) at Day 0 and at Month 3
Description: The antibodies against BPT assessed were against pertussis toxoid (anti-PT), against filamentous haemagglutinin (anti-FHA), and against pertactin (anti-PRN). Concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs), in ELISA units per milliliter (EL.U/mL). The cut-off of the assay was the seropositivity cut-off value of greater than or equal to (>=) 5 EL.U/mL. The table shows results for study groups pooled by primary vaccine administered (RTS,S vs Engerix -B)
Time Frame: At Day 0 and at Month 3 (one month post Dose 3 of Infanrix-Hib)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- Engerix B Group: Subjects in this group were subjects from the Engerix B Regimen A and Engerix B Regimen B groups were administered Engerix B as a 3-dose primary vaccination course, at Weeks 0, 4 and 8, followed by a booster dose, at Month 50. Subjects in this group were also administered, according to varied schedules, depending on the vaccination regimen they were allocated too in their respective group, doses Infanrix-Hib, Polio Sabin, Rotarix, Synflorix, Rotarix and of vaccines against yellow fever and against measles. Engerix B was administered intramuscularly (IM) in the left anterolateral thigh, Infanrix-Hib IM in the right deltoid, Synflorix IM in the right anterolateral thigh, and Rotarix and Polio Sabin orally. The measles and yellow fever vaccines were administered IM in the deltoid.
Arm/Group | RTS,S Group | Engerix B Group
Number analyzed (Participants) | 401 | 253
EL.U/mL
  Anti-PT - At Day 0 | 3.8 [3.6 to 4.1] | 4.3 [3.9 to 4.8]
  Anti-PT - At Month 3: number analyzed (Participants) | 387 | 247
  Anti-PT - At Month 3 | 105.9 [99.2 to 113.1] | 114.2 [104.8 to 124.5]
  Anti-FHA - At Day 0: number analyzed (Participants) | 399 | 253
  Anti-FHA - At Day 0 | 13.9 [12.7 to 15.2] | 15.7 [14.1 to 17.5]
  Anti-FHA - At Month 3: number analyzed (Participants) | 386 | 247
  Anti-FHA - At Month 3 | 271.1 [252.8 to 290.8] | 292.9 [268.9 to 319.1]
  Anti-PRN - At Day 0 | 3.2 [3.0 to 3.4] | 3.2 [3.0 to 3.5]
  Anti-PRN - At Month 3: number analyzed (Participants) | 387 | 247
  Anti-PRN - At Month 3 | 164.1 [153.6 to 175.3] | 179.7 [164.4 to 196.5]
Statistical Analysis 1: Comparison: RTS,S Group vs Engerix B Group; To demonstrate the non-inferiority of antibody response to the acellular B pertussis antigen, pertussis toxoid, (PT) of the DTPa/Hib vaccine when co-administered with RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — Criteria for non-inferiority: one month post Dose 3, upper limit (UL) of the 2-sided 95% confidence interval (CI) on the GMC ratios of anti-PT, anti-FHA, anti-PRN antibody concentrations, is below a limit of 2 for the DTPa/Hib vaccine when co-administered with versus without RTS,S/AS01E; ANOVA; GMC ratio = 1.08, 95% CI 2-sided [0.97 to 1.20]
Statistical Analysis 2: Comparison: RTS,S Group vs Engerix B Group; To demonstrate the non-inferiority of antibody response to the acellular B pertussis antigen, filamentous haemagglutinin (FHA), of the DTPa/Hib vaccine when co-administered with RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; ANOVA; GMC ratio = 1.08, 95% CI 2-sided [0.97 to 1.21]
Statistical Analysis 3: Comparison: RTS,S Group vs Engerix B Group; To demonstrate the non-inferiority of antibody response to the acellular B pertussis antigen, pertactin (anti-PRN), of the DTPa/Hib vaccine when co-administered with RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — [test comment as in outcome 18, analysis 1]; ANOVA; GMC ratio = 1.10, 95% CI 2-sided [0.98 to 1.22]

19. Secondary Outcome: Anti-Rotavirus (Anti-RV) Antibody Concentrations
Description: Anti-Rotavirus (anti-RV) antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs). The cut-off of the assay was the seropositive cut-off value of greater than or equal to (>=) 20 units per milliliter (U/mL). This outcome measure was assessed in subjects who were administered Rotarix as part of an EPI regimen, with and without RTS,S vaccine co-administration. This outcome concerns the subjects who received the RTS,S or Engerix-B vaccine co-administered with Rotarix. Results presented are for the study groups pooled by RTS,S or Engerix-B vaccine co-administration, that is, for the RTS,S Regimen B and Engerix-B Regimen B groups.
Time Frame: At Month 3, aka one month post Dose 2 of Rotarix
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | RTS,S Regimen B Group | Engerix B Regimen B Group
Number analyzed (Participants) | 120 | 116
U/mL | 24.9 [19.3 to 32.0] | 27.6 [20.8 to 36.5]
Statistical Analysis 1: Comparison: RTS,S Regimen B Group vs Engerix B Regimen B Group; To demonstrate the non-inferiority of antibody response to the rotavirus vaccine when co-administered with versus without RTS,S/AS01E as part of an EPI regimen; Test type: Non-Inferiority — Criteria for non-inferiority: one month post Dose 2, upper limit (UL) of the 2-sided 95% confidence interval (CI) on the geometric mean concentrations (GMC) ratios of rotavirus antibodies (IgA) concentrations is below 2 for the rotavirus vaccine when co-administered with versus without RTS,S/AS01E; ANOVA; GMC ratio = 1.11, 95% CI 2-sided [0.76 to 1.61]

20. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling at the site of injection. All solicited local symptoms assessed were considered by the investigator as causally related to the study vaccination. Analysis for this outcome was performed solely for the 7-days follow-up periods following the primary vaccination with RTS,S vaccine or Engerix-B (at Day 0, and Months 1 and 2). Data presented are those for any occurrence of the assessed solicited local symptoms, that is, the occurrences of these symptoms regardless of their intensity grade.
Time Frame: Within the 7-day follow-up period (Days 0-6) after administration of Dose (D) 1, 2 and 3, respectively, with RTS,S or Engerix-B vaccine
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had their symptom sheets filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants
  Pain - Post D1 | 41 | 28 | 31 | 29 | 15
  Pain - Post D2: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Pain - Post D2 | 30 | 14 | 21 | 24 | 9
  Pain - Post D3: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Pain - Post D3 | 14 | 10 | 14 | 18 | 7
  Redness - Post D1 | 1 | 0 | 2 | 5 | 1
  Redness - Post D2: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Redness - Post D2 | 5 | 1 | 2 | 3 | 0
  Redness - Post D3: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Redness - Post D3 | 3 | 0 | 1 | 3 | 0
  Swelling - Post D1 | 5 | 2 | 6 | 10 | 4
  Swelling - Post D2: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Swelling - Post D2 | 8 | 3 | 4 | 9 | 4
  Swelling - Post D3: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Swelling - Post D3 | 7 | 2 | 6 | 11 | 3

21. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fever, irritability/fussiness, drowsiness, and loss of appetite. Fever was defined as axillary temperature higher than (>) 37.5 degrees Celsius (°C). Analysis for this outcome was performed solely for the 7-days follow-up periods following the primary vaccination with RTS,S vaccine or Engerix-B (at Day 0, and Months 1 and 2). Data presented are those for any occurrence of the assessed solicited general symptoms, that is, the occurrences of these symptoms regardless of their intensity grade or relationship to vaccination.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants
  Fever - D1 | 44 | 20 | 16 | 23 | 13
  Fever - D2: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Fever - D2 | 30 | 14 | 18 | 20 | 5
  Fever - D3: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Fever - D3 | 38 | 20 | 26 | 16 | 12
  Irritability - D1 | 15 | 11 | 11 | 9 | 5
  Irritability - D2: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Irritability - D2 | 13 | 7 | 12 | 10 | 0
  Irritability - D3: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Irritability - D3 | 5 | 3 | 10 | 6 | 1
  Drowsiness - D1 | 2 | 1 | 3 | 3 | 0
  Drowsiness - D2: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Drowsiness - D2 | 5 | 1 | 1 | 3 | 0
  Drowsiness - D3: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Drowsiness - D3 | 3 | 0 | 2 | 1 | 0
  Loss of appetite - D1 | 4 | 1 | 2 | 4 | 0
  Loss of appetite - D2: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Loss of appetite - D2 | 3 | 1 | 1 | 3 | 0
  Loss of appetite - D3: number analyzed (Participants) | 141 | 126 | 141 | 141 | 123
  Loss of appetite - D3 | 2 | 0 | 1 | 1 | 1

22. Secondary Outcome: Number of Subjects With Potential Immune Mediated Disorders (pIMDs) From Day 0 to Month 8
Description: A potential immune mediated disorder (pIMD) was defined as an event about which concerns arose that vaccination may have interfered with immunological self-tolerance of the subjects. IMDs assessed included among others neuroinflammatory disorders (such as optic neuritis, multiple sclerosis, or encephalitis), musculoskeletal disorders (such as cutaneous lupus, rheumatoid arthritis, juvenile arthritis, or psoriatic arthropathy), gastrointestinal disorders (ulcerative colitis and ulcerative proctitis, celiac disease), metabolic diseases (such as autoimmune thyroiditis, or diabetes Mellitus Type 1, Addison's disease), skin disorders (such as psoriasis or vitiligo), and other disorders such as vasculitis, pernicious anemia, or, sarcoidosis.
Time Frame: From Day 0 to Month 8
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Subjects With Potential Immune Mediated Disorders (pIMDs) From Day 0 to Month 26
Description: as for outcome 22
Time Frame: From Day 0 to Month 26
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects With Potential Immune Mediated Disorders (pIMDs) From Day 0 up to Study End (Month 51)
Description: as for outcome 22
Time Frame: From Day 0 up to Study End (Month 51)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 30-day follow-up periods (Days 0-29) after vaccination with RTS,S vaccine or Engerix-B
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants | 121 | 115 | 120 | 120 | 105

26. Secondary Outcome: Number of Subjects With Any and Fatal Serious Adverse Events (SAEs) Within the 30-day Follow-up Periods (Days 0-29)
Description: A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or a reported adverse event of specific interest such as seizures occurring within a 30-day period of vaccination, immune-mediated disorders, and specific autoimmune diseases. A fatal SAE was defined as a SAE resulting in the death of the study subject.
Time Frame: Within the 30-day follow-up periods (Days 0-29) after vaccination with RTS,S vaccine or Engerix-B
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants
  Subject with SAE(s) | 1 | 3 | 3 | 1 | 3
  Subjects with fatal SAE(s) | 1 | 0 | 1 | 0 | 0

27. Secondary Outcome: Number of Subjects With Any and Fatal Serious Adverse Events (SAEs) From Day 0 to Month 8
Description: as for outcome 26
Time Frame: From Day 0 to Month 8
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants
  Subjects with SAE(s) | 1 | 7 | 7 | 3 | 5
  Subjects with fatal SAE(s) | 1 | 2 | 2 | 0 | 0

28. Secondary Outcome: Number of Subjects With Any and Fatal Serious Adverse Events (SAEs) From Day 0 to Month 26
Description: as for outcome 26
Time Frame: From Day 0 to Month 26
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants
  Any SAEs - At Month 26 | 1 | 8 | 7 | 6 | 6
  Fatal SAEs - At Month 26 | 1 | 3 | 2 | 2 | 1

29. Secondary Outcome: Number of Subjects With Any, Fatal and Related Serious Adverse Events (SAEs) From Day 0 up to Study End (Month 51)
Description: A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or a reported adverse event of specific interest such as seizures occurring within a 30-day period of vaccination, immune-mediated disorders, and specific autoimmune diseases. A fatal SAE was defined as a SAE resulting in the death of the study subject. A related SAE was defined as a SAE assessed by the investigator as being causally related to vaccination.
Time Frame: From Day 0 up to Study End (Month 51)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
Number analyzed (Participants) | 142 | 142 | 141 | 141 | 139
Participants
  Any SAEs | 3 | 10 | 9 | 6 | 6
  Fatal SAEs | 3 | 5 | 4 | 2 | 1
  Related SAEs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local, general symptoms and unsolicited AEs: within the 30-day periods after primary co-administration vaccination. SAEs: during the entire study period (Month 0 to Month 51).
Arm/Group | RTS,S Regimen A Group | RTS,S Regimen B Group | RTS,S Regimen C Group | Engerix B Regimen A Group | Engerix B Regimen B Group
All-Cause Mortality (participants affected / at risk) | 3/142 | 5/142 | 4/141 | 2/141 | 1/139
Serious Adverse Events (participants affected / at risk) | 3/142 | 10/142 | 9/141 | 6/141 | 6/139
Other Adverse Events (participants affected / at risk) | 135/142 | 129/142 | 132/141 | 135/141 | 119/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTS,S Regimen A Group (N=142) | RTS,S Regimen B Group (N=142) | RTS,S Regimen C Group (N=141) | Engerix B Regimen A Group (N=141) | Engerix B Regimen B Group (N=139)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Intravascular haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Salmonella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Trichomoniasis intestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTS,S Regimen A Group (N=142) | RTS,S Regimen B Group (N=142) | RTS,S Regimen C Group (N=141) | Engerix B Regimen A Group (N=141) | Engerix B Regimen B Group (N=139)
Somnolence (Nervous system disorders) | 8 (10) | 2 (2) | 5 (6) | 5 (7) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Abscess (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anal fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 8 (9) | 5 (5) | 5 (5) | 4 (4) | 4 (4)
Bronchitis (Infections and infestations) | 36 (47) | 33 (35) | 28 (35) | 28 (31) | 29 (37)
Bullous impetigo (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 8 (8) | 10 (10) | 11 (12) | 9 (10) | 7 (7)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (9) | 2 (2) | 4 (4) | 5 (8) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 19 (19) | 8 (8) | 20 (20) | 12 (13) | 6 (6)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 3 (3) | 3 (3) | 5 (5) | 3 (3) | 4 (4)
Fungal skin infection (Infections and infestations) | 1 (1) | 7 (7) | 6 (6) | 12 (12) | 4 (4)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 42 (55) | 47 (58) | 51 (71) | 43 (57) | 38 (47)
Gastrointestinal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 28 (33) | 18 (21) | 27 (33) | 19 (25) | 5 (6)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 44 (50) | 44 (54) | 39 (46) | 49 (52) | 44 (53)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Oral candidiasis (Infections and infestations) | 5 (5) | 3 (3) | 3 (3) | 4 (4) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 11 (11) | 12 (13) | 6 (6) | 15 (19) | 10 (11)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 55 (85) | 40 (52) | 47 (66) | 48 (71) | 25 (32)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 23 (24) | 13 (15) | 15 (19) | 15 (18) | 17 (18)
Pneumonia (Infections and infestations) | 5 (5) | 14 (15) | 4 (4) | 11 (11) | 2 (2)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 5 (7) | 7 (7) | 5 (5) | 6 (7) | 3 (3)
Pyrexia (General disorders) | 81 (116) | 49 (56) | 50 (66) | 55 (65) | 34 (37)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 10 (10) | 14 (16) | 15 (18) | 12 (13) | 10 (11)
Respiratory tract malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 32 (37) | 35 (41) | 33 (41) | 31 (36) | 31 (36)
Skin bacterial infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 17 (20) | 7 (7) | 14 (16) | 23 (30) | 10 (11)
Tinea infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (18) | 8 (9) | 12 (15) | 8 (9) | 7 (10)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Visceral larva migrans (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol (2014-05-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT01345240/Prot_000.pdf